CLINICAL TRIAL: NCT00597090
Title: The Role of Genetic Polymorphisms in Innate Immune Response Genes in Susceptibility to Infections
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Papanicolaou, Genovefa, MD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 03-017
Record Dates: First submitted 2008-01-08; First posted 2008-01-17 (Estimated); Last update posted 2011-01-20 (Estimated); Status verified 2011-01

CONDITIONS: Infections
Keywords: Infections; lymphoma
MeSH Terms: conditions — Infections; Lymphoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will genotype the genes of innate immune receptors to identify genetic polymorphisms associated with higher frequency of invasive infections or susceptibility to lymphoma. All specimens will be processed in the Infectious Diseases Laboratory at MSKCC. RNA will be extracted from peripheral blood mononuclear cells (PBMCs). Genotyping will be done from genomic DNA or from cDNA generated from RNA by RT-PCR. Cell lines will be created from PBMCs and will be analyzed in functional assays for responses to bacterial and fungal products (cytokine secretion, upregulation of cell surface molecules). All patient samples including genomic DNA, RNA, cDNA and cell lines will be banked in the Infectious Disease laboratory at MSKCC.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
The purpose of this study is to better understand genetic susceptibility to infections and the interactions of specific genetic polymorphisms of innate immune receptors with microbial and fungal organisms.

The goals of this study are:

1. Find out if some people are more likely to get severe infections, than others. To do this we will compare patients with leukemia who develop severe infections to patients who do not develop infections.
2. Find out if some people are more likely to develop lymphoma than others. To do this we will compare patients with lymphoma to people without lymphoma who are of the same sex and similar age and ethnic background to the patients with lymphoma.

DETAILED DESCRIPTION:
A small number of patients will develop severe infection after chemotherapy or after allogeneic bone marrow transplantation. The ability of patients with leukemia or bone marrow transplantation to fight infections is decreased. One reason is that chemotherapy transiently destroys the type of white blood cells called neutrophils. Neutrophils are the first line of defense of our body against infections. Bone marrow transplant patients may be receiving edications to prevent graft versus host disease. Such medications may decrease the ability of the body to fight infections.

People respond to infections in different ways. Some may be born with genes that make them more likely to get certain types of infections. Specific genes may affect the response to different microbes (pathogens). We want to find out which genes have normal changes in them and lead to different responses to infections. We also want to find out how the ability to fight infections is related to the way these genes work.

Responses to infection are controlled by our immune system. Changes in genes of the immune system that may alter control of infection may make people more susceptible to some types of lymphoma The goals of this study are:

1. Find out if some people are more likely to get severe infections, than others. To do this we will compare patients with leukemia who develop severe infections to patients who do not develop infections.
2. Find out if some people are more likely to develop lymphoma than others. To do this we will compare patients with lymphoma to people without lymphoma who are of the same sex and similar age and ethnic background to the patients with lymphoma.

The purpose of this study is to better understand genetic susceptibility to infections and the interactions of specific genetic polymorphisms of innate immune receptors with microbial and fungal organisms.

To accomplish this, blood specimens from patients with acute myeloid leukemia, RAEB, RAEBT or acute lymphocytic leukemia, follicular or mantle cell lymphoma or recipients of allogeneic hematopoietic stem cell transplants (HSCT) will be collected. We will genotype the genes of innate immune receptors to identify genetic polymorphisms associated with higher frequency of invasive infections or susceptibility to lymphoma. All specimens will be processed in the Infectious Diseases Laboratory at MSKCC. RNA will be extracted from peripheral blood mononuclear cells (PBMCs). Genotyping will be done from genomic DNA or from cDNA generated from RNA by RT-PCR. Cell lines will be created from PBMCs and will be analyzed in functional assays for responses to bacterial and fungal products (cytokine secretion, upregulation of cell surface molecules). All patient samples including genomic DNA, RNA, cDNA and cell lines will be banked in the Infectious Disease laboratory at MSKCC.

In order to perform this study, patients diagnosed with acute leukemia will be asked to provide blood, and permission to review the medical charts. We will collect (removed prospectively) data regarding risk factors for infections, diagnosis of infections, response to treatment and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Subject must either:

  1. Have histologically confirmed acute myeloid leukemia (AML), acute lymphocytic leukemia (ALL), follicular or mantle cell lymphoma RA-EB, RAEB-T newly diagnosed at first or second remission AND are going to receive or have received myelosuppressive chemotherapy; OR
  2. Will receive or have received allogeneic HSCT for hematologic malignancy.
* Subject has signed informed consent before entering the study.

Participation of children: For subjects under the age of 18, we will obtain the subject's and their parents' approval to enroll them.

Exclusion Criteria:

* Subject has been diagnosed with leukemia other than acute myeloid leukemia RA-EB or RAEB-T or acute lymphocytic.
* Subject is not going to receive chemotherapy or has not received chemotherapy.
* Subject will undergo/had undergone HSCT for disease other than hematologic malignancy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population for this study is composed of patients with leukemia. It is projected that the marginal probability of an allelic variant in the TLR and an infection is 0.12 and 0.30 respectively in this patient population.
Sampling Method: Probability Sample
Enrollment: 319 (Actual)
Dates: Start 2003-02; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Risk for developing infection or lymphoma due to allelic variation in genes of immune system that specialize in pathogen recognition compared to absence of allelic variation. | 6 years

SECONDARY OUTCOMES:
Risk for developing infectns due to somatic mutatns/polymorphisms in genes involved in signaling pathways downstream of receptors of immune recognitn.Characterize in vitro diff in functional responses to pathogens among genetic variants. | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Genovefa Papanicolaou, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org